CLINICAL TRIAL: NCT05007678
Title: Targeting de Novo Pyrimidine Biosynthesis by Leflunomide as a Novel Concept for the Treatment of Corona Virus Disease 2019 (COVID-19)
Brief Title: Targeting de Novo Pyrimidine Biosynthesis by Leflunomide for the Treatment of COVID-19 Virus Disease
Acronym: DEFEAT-COVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ashford and St. Peter's Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020ZC01
Record Dates: First submitted 2021-07-16; First posted 2021-08-16 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: COVID-19; Leflunomide; Acute emergency care
MeSH Terms: conditions — COVID-19 | interventions — Leflunomide

STUDY DESIGN:
Intervention Model Description: Randomised
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): The usual care will be offered as per current advice on management of hospitalised patients.
- leflunomide (Active Comparator): Patients admitted to the hospital COVID-19 positive and within 2 weeks of symptoms' onset will be treated with loading dose of 100 mg leflunomide for 3 days, followed by 20 mg once daily. Participants with ALT/AST levels 2 times above upper limits of normal reference range will receive 10mg instead of 20mg.
  Interventions: Drug: leflunomide

INTERVENTIONS:
Drug: leflunomide — leflunomide administered orally; daily loading dose of 100mg for 3 days, followed by a daily maintenance dose 10-20mg daily, to a total course of 10 days
  Arms: leflunomide

SUMMARY:
The global COVID-19 pandemic has caused unprecedented strain on health care services around the world.The absence of specific anti-viral medications to treat the underlying infection led to a proliferation of clinical studies and trials aimed at re-purposing existing medications.

Human dihydroorotate dehydrogenase (DHODH) is vital enzyme utilised by viruses to replicate in the host cell. Leflunomide, a drug that is already licenced to treat rheumatoid arthritis, is a potent inhibitor of the enzyme DHODH. Importantly, this drug has dual anti-viral and anti-inflammatory properties so it targets viral replication and suppresses host inflammatory response which plays a role at more progressive stages of infection.

DEFEAT-COVID is a multi-site, international, interventional, pragmatic, parallel group design, open label, randomised CTIMP with a pilot phase that will allow to adapt procedures and assessments if required.

A phase III clinical trial of leflunomide for treating COVID-19 has been registered in China, Registration number: ChiCTR2000030058). The current proposal extends the original clinical study of leflunomide in China (People's Hospital of Wuhan University) to the UK through a structured collaboration.

DETAILED DESCRIPTION:
Leflunomide is a potent inhibitor of the enzyme DHODH and is already licenced to treat rheumatoid arthritis. Importantly, this drug has dual anti-viral and anti-inflammatory properties which is advantageous in COVID-19 infected patients, as more progressive stages of the disease involve augmented responses from the host inflammatory mechanisms leading to serious complications and death.

Based on the current understanding of the pathogenesis of COVID-19 infection and its spectrum of clinical manifestation it is evident that a significant proportion of those infected develop pneumonia, systemic inflammatory response and cardiovascular complications with high morbidity and mortality. The progression from initial mild symptoms (usually fever, fatigue and cough) to severe pneumonia requiring oxygen support or mechanical ventilation often takes one to two weeks after the onset of symptoms. The progression leading to a such deterioration is thought to be related to the kinetics of viral replication culminating in an exaggerated surge in inflammatory mediator release, called "cytokine storm".

Host-targeting antiviral (HTA) strategies have many advantages to fight against a broad spectrum of viruses compared to direct-acting antiviral drugs. These include blocking the viral replication and overcoming the potential of viral mutagenesis simultaneously.

Concept The quest for optimal HTA strategies enabled the investigators to identify a crucial enzyme called human dihydroorotate dehydrogenase (DHODH) that limits pyrimidine synthesis. This is a vital metabolic process utilised by viruses for replication.

In preclinical models of cell and animal infection by SARS-CoV-2 the DHODH inhibitors exhibited multiple actions including attenuation of viral genome replication, suppression of the inflammatory reaction and the release of pro-inflammatory cytokines and chemokine. These drugs also offered protection against mortality in mice when administered at later stages of infection when direct acting antivirals offered no survival benefit. The hypothesis is that DHODH inhibitors may have the advantage in treatment of COVID-19 disease even at its advanced stage compared to the drugs with either standalone anti-viral or anti-inflammatory properties.

To this end, collaborators in China have conducted a pilot study in COVID-19 patients in Wuhan, the epicentre of China COVID-19 outbreak, with moderate clinical symptoms. This study has demonstrated feasibility with a favourable clinical outcome and good safety profile within the leflunomide treatment arm. Patients receiving leflunomide had a shorter clinical recovery time and a reduction in clinical inflammatory biomarkers with no side effects observed.

Leflunomide This is an immunosuppressive agent whose efficacy and safety profiles are well established in treatment of rheumatoid arthritis. In 76 000 patients treated with leflunomide there were 16 potential cases of pancytopenia and 9 cases of serious skin reactions. It has few GI side effects including derangement in liver function, associated with long-term use.

The recommended dosage of leflunomide in COVID-19 is a loading dose of 100 mg/day for 3 days, followed by 10-20 mg once daily depending on liver functions (patients with ALT/AST levels above upper limits of normal (ULN) reference range will have 10mg instead of 20mg). This regimen is routinely used in the treatment of rheumatoid arthritis providing effective blood concentration and few adverse reactions.

Leflunomide not only inhibits SARS-CoV-2 viral genome replication but also suppresses the release of pro-inflammatory cytokines and chemokines, suggesting its potential advantage in treating the SARS-CoV-2-induced COVID-19 disease compared to the drugs with standalone anti-viral or anti-inflammatory properties.

Rapidly replicating viruses rely on the de novo pyrimidines biosynthesis to acquire sufficient pyrimidines for genome replication. By inhibiting the host target DHODH, leflunomide can block the de novo pyrimidine biosynthesis by inhibiting the rate limiting step for the viral nucleic acid (DNA and RNA) replication process. The in-vitro data have shown it to be effective against a broad-spectrum of viruses.

Objectives and Outcome Measures/ Endpoints The main trial objective is to evaluate the clinical efficacy and safety of 10 days oral leflunomide treatment starting within 2 weeks of moderate to critical illness symptoms' onset in patients with confirmed COVID-19 infection.

Additionally, the study will evaluate the impact of leflunomide on:

1. the rate of viral clearance
2. the extent of lung injury, based on CT imaging and on the need of invasive/non-invasive ventilation and respiratory support.
3. myocardial, kidney, and liver function based on the need for inotropic/vasoactive and mechanical support and renal replacement therapy.
4. assessment of respiratory, myocardial and kidney injury assessed by standardised physiological and biomarker criteria including emerging molecular and inflammatory footprints of COVID-19 disease Based on the measured variables models to predict the severity of the disease as well as clinical outcomes will be built.

Trial Design The World Health Organisation (WHO) "master protocol" i.e. the R&D blueprint Therapeutic Trial Synopsis for COVID-19 was taken into account when designing the trial. This is illustrated in how the trial is conducted i.e. i) using a 2 stage approach of including a pilot phase before a main trial, ii) target population, ii) participant eligibility, iv) primary and secondary outcomes / endpoints, and v) the trial assessments needed to meet the objectives of ensuring clinical benefit and patient safety of the new therapy being investigated.

The number of patient visits and assessments conducted are kept to a minimum but sufficient to address both the immediate and long term risk to public health. This takes into account conventional standard operating procedures, Good Clinical Practice (GCP), national and international clinical trial regulations.

DEFEAT-COVID is a multi-site, international, interventional, pragmatic, parallel group design, open label, randomised CTIMP with a pilot phase that will allow us to adapt procedures and assessments if required.

Trial Setting The study is primarily conducted at secondary and tertiary healthcare settings in England and India. At each local clinical centre (LCC), the principal investigator (P)I will be responsible for trial activities but much of the work will be carried out by medical staff providing care to patients with COVID-19 within the hospital and by hospital research nurses, medical students and other staff when delegated and with appropriate education, training, and experience.

The landscape of the COVID infection in London and other regions in the UK is being monitored. Additional sites will be invited to contribute to the trial upon recommendation by the Steering and Trial Management Committees taking into consideration of developing national hotspots, second wave of the pandemic etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years,
2. Patients with onset of symptoms >15 days,
3. Laboratory (RT-PCR) confirmed infection with 2019-nCoV.

Exclusion Criteria:

1. Pregnant or breast feeding,
2. On specific monoclonal antibodies, or other drug trial treatment for COVID-19 within one week prior to study enrolment,
3. Liver function tests >2 fold of upper limits of normal (ULN) reference levels of the respective testing assay,
4. Patients with known hypersensitivity to leflunomide,
5. Patients with severe immunodeficiency syndrome and hypoalbuminaemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement | 28 days from randomisation
  TTCI is defined as the time (in days) from initiation of trial treatment (for participants in the treatment arm), or day of randomisation (for participants in the control arm), until the first occurrence of;
  1. an improvement of two points on a seven-category ordinal scale of clinical status categories.All surviving patients who have not reached any TTCI ordinal level by Day 28 will be right-censored at that point.
  2. live discharge from hospital.
Incidence of adverse events | 28 days from randomisation
  All adverse events within 28 days will be recorded and incidence of serious adverse events (SAEs) and Grade 3 and 4 adverse events (AEs)* will be reported.
  *Grade 3 adverse events: Severe or medically significant but not immediately life-threatening; or hospitalisation or prolongation of hospitalisation indicated; or disabling; or limiting self-care activity of daily living. Grade 4 Life-threatening consequences; urgent intervention indicated.

SECONDARY OUTCOMES:
Changes in virological load over time | Days 0/1, 7,11 and 15 days post randomisation
  Comparing changes in virological load at predefined time periods by comparing proportions of SARS-CoV-2 negativity by RT-PCR and changes in viral load in upper respiratory tract specimens.
Time to hospital discharge | Daily assessments during hospitalisation up to 28 days or discharge
  Number of days from randomisation to discharge
All-cause mortality | From randomisation to the event within 28 days
  Recorded incidence of mortality due to any cause
Duration of intensive care stay | From randomisation to 28 days or discharge
  Time from admission to ITU to discharge to another care environment will be recorded for each patient, noting that the start of this period may ante-date the time of randomisation.
Duration of invasive and non-invasive ventilation | From randomisation to discharge or 28 days
  Time from initiation to withdrawal of mechanical ventilation will be recorded, subdivided by whether the ventilation was invasive.
Incidence of re-intubation | From randomisation to 28 days or discharge
  The proportion of patients requiring re-intubation following a decision to extubate
Incidence of tracheostomy | From randomisation to 28 days or discharge
  The proportion of patients requiring tracheostomy
Degree of acute lung injury | At baseline, 15 and 28 days or discharge
  Proportions of patients with mild, moderate and severe lung impairment based on Berlin definition
Evaluation of surrogate of inflammation and lung recovery | Daily measurements from randomisation to discharge or 28 days
  Ratios of arterial and peripheral oxygen saturation divided by fraction of inspired oxygen:
  * P/F ratio, (i.e. arterial pO2 divided by the FIO2)
  * S/F ratio, (i.e. oxygen saturation divided by the FIO2)
Incidence of inotropic/vasoactive support | From randomisation to discharge or 28 days
  The proportion of patients needing inotropic/vasoactive support
Incidence of acute kidney injury | From randomisation to discharge or 28 days
  Proportion of patients diagnosed with acute kidney injury by the KDIGO criteria
Need for renal replacement therapy | From randomisation to discharge or 28 days
  Proportion of patients needing renal replacement therapy
Characterisation of biomarkers including high sensitivity CRP, ferritin, procalcitonin, troponin, BNP, creatinine and kidney biomarkers. | Daily measurements during hospitalisation to 28 days or discharge
  Measurements of these markers will be collected daily
Changes in cytokine profile including pro- and anti-inflammatory cytokines | Days 0, 1, 3 and 11
  Measurements for each of the cytokines will be collected at predetermined time points.

OTHER OUTCOMES:
Evaluation of patient reported symptoms in follow up | 30 and 90 days after discharge
  Completion of questionnaires to examine persistence of any COVID-19 related symptoms of COVID-19 persisted

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Chen, CI, Study Chair — Ashford and St Peters Hospital NHS Foundation Trust; Isaac John, Study Director — Ashford and St Peters Hospital NHS Foundation Trust; Sharma Shashank, PI, Principal Investigator — Ashford and St Peters Hospital NHS Foundation Trust
Locations (1):
- Ashford and St Peters Hospital NHS Foundation Trust, Chertsey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the data supporting the results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 2 years from publication of the main results
Access Criteria: The anonymized data may be made available upon request following approval from the Trial Management Group and the Sponsor.

REFERENCES:
- [Derived] Kralj-Hans I, Li K, Wesek A, Lamorgese A, Omar F, Ranasinghe K, McGee M, Brack K, Li S, Aggarwal R, Bulle A, Kodre A, Sharma S, Fluck D, John I, Sharma P, Belsey JD, Li L, Seshasai SRK, Li HL, Marczin N, Chen Z; DEFEAT-COVID Investigators. Leflunomide treatment for patients hospitalised with COVID-19: DEFEAT-COVID randomised controlled trial. BMJ Open. 2023 Apr 13;13(4):e068179. doi: 10.1136/bmjopen-2022-068179. PMID 37055207